CLINICAL TRIAL: NCT03503214
Title: Changes in Acid-base Variables Induced by Acute Variations in Partial Pressure of Carbon Dioxide in Whole Blood and Isolated Plasma of Septic Critically Ill Patients and Healthy Volunteers: an In-vitro Study
Brief Title: Non Carbonic Buffer Power of Critical Ill Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: Buffer power
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-03

CONDITIONS: Acid-Base Imbalance; Respiratory Acidosis; Respiratory Alkalosis
Keywords: Acid-base equilibrium; Stewart's approach; In vitro study; Respiratory acid-base derangements
MeSH Terms: conditions — Acid-Base Imbalance; Acidosis, Respiratory; Alkalosis, Respiratory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic patients: Patients with sepsis or septic shock according to the SEPSIS-III (Singer M Jama 2016) admitted to the general Intensive Care Unit
  Interventions: Diagnostic Test: In vitro determination of non-carbonic buffer power; Diagnostic Test: Classic description of acid-base status
- Healthy volunteers: Subjects without known respiratory, cardiovascular, hepatic, renal or hematologic diseases.
  Interventions: Diagnostic Test: In vitro determination of non-carbonic buffer power; Diagnostic Test: Classic description of acid-base status

INTERVENTIONS:
Diagnostic Test: In vitro determination of non-carbonic buffer power — In vitro measurement of the non-carbonic buffer power by the means of equilibration of whole blood and isolated plasma with gas mixtures containing different concentrations of carbon dioxide
Diagnostic Test: Classic description of acid-base status — Measurement of plasma electrolytes, hemoglobin concentration, albumin and phosphates to compute acid-base variables according to Stewart's approach.

SUMMARY:
Alterations of acid-base equilibrium are very common in critically ill patients and understanding their pathophysiology can be important to improve clinical treatment.

The human organism is protected against acid-base disorders by several compensatory mechanisms that minimize pH variations in case of blood variations in carbon dioxide content. The aim of the present study is to quantify the buffer power, i.e. the capacity to limit pH variations in response to carbon dioxide changes, in critically ill septic patients and compare these results with data collected from healthy volunteers.

DETAILED DESCRIPTION:
Alterations of acid-base equilibrium are very common in critically ill patients and understanding their pathophysiology can be important to improve clinical treatment.

The human body is protected against acid-base disorders by several compensatory mechanisms that minimize pH variations in response to acid-base derangements.

The present study focuses on the acute compensatory mechanisms of respiratory acid-base derangements, i.e., respiratory acidosis and respiratory alkalosis. In this case the non-carbonic buffers are constituted by albumin and phosphates in plasma, with the addition of hemoglobin in whole blood.

Aim of the present in-vitro study is to measure the buffer power of non-carbonic weak acids contained in whole blood and isolated plasma, assess the relative contribution of red blood cells and plasma proteins and perform a comparison between septic patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Septic patients and healthy volunteers

Exclusion Criteria:

* age < 18 years and pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock admitted to the ICU will be enrolled. Furthermore, healthy volunteers recruited from ICU staff members and relatives will be enrolled as control group.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Non-carbonic buffer power | 1 day
  Non-carbonic buffer power (beta) of whole blood and isolated plasma [expressed as variations in bicarbonate concentration divided by variations in pH).

SECONDARY OUTCOMES:
Strong Ion Difference variations induced by carbon dioxide | 1 day
  Variations in Strong Ion Difference of whole blood and plasma [expressed in milliequivalents per Liter], induced by acute in vitro changes of carbon dioxide
Bicarbonate Variations induced by carbon dioxide | 1 day
  Variations in bicarbonate concentration of whole blood and plasma [expressed in milliequivalents per Liter], induced by acute in vitro changes of carbon dioxide
Oxidized albumin | 1 day
  Oxidized albumin [expressed as percentage of total albumin concentration]
Correlation between hematocrit values and Strong Ion Difference variations | 1 day
  Correlation between hematocrit [expressed as percentage] values and Strong Ion Difference variations [expressed in mEq/L] induced by acute in vitro changes of Carbon Dioxide.
  Acute variations in partial pressure of carbon dioxide cause changes in Strong Ion Difference. The hypothesis is that the magnitude of Strong Ion Difference variations correlate to the hematocrit, being the red blood cell the major source of electrolytes. The higher the hematocrit, the higher the possible change in Strong Ion Difference induced by acute variations in partial pressure of carbon dioxide.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Langer, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano; Antonio Pesenti, MD, Study Director — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano; Giacomo Grasselli, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano
Locations (1):
- IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy